CLINICAL TRIAL: NCT01069094
Title: A Single Dose lead-in PK Followed by a Randomized, Double-blinded, Controlled, Multiple Dose Study of the Selective Progesterone Receptor Modulator Progenta (CDB-4124) in Pre-menopausal Women With Symptomatic Leiomyomata
Brief Title: A Study of Progenta (CDB-4124) in Pre-menopausal Women With Symptomatic Leiomyomata
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZN-001
Record Dates: First submitted 2010-02-12; First posted 2010-02-17 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2014-06

CONDITIONS: Uterine Leiomyomata
Keywords: Uterine fibroids
MeSH Terms: conditions — Myofibroma; Leiomyoma | interventions — telapristone acetate; Leuprolide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- progenta 12.5 mg (Experimental): Progenta (CDB-4124) 12.5 mg capsule
  Interventions: Drug: Progenta
- progenta 25 mg (Experimental): Progenta (CDB-4124) 25 mg capsule
  Interventions: Drug: Progenta
- progenta 50 mg (Experimental): Progenta (CDB-4124) 50 mg capsule
  Interventions: Drug: Progenta
- Lucron Depot (Active Comparator): Lucron Depot, Leuprolide acetate for depot suspension
  Interventions: Drug: Lucron Depot
- placebo (Placebo Comparator): Placebo capsule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Progenta — 12.5 mg, administered as a once daily oral dose for 90 days.
  Other Names: CDB-4124; Telapristone acetate
  Arms: progenta 12.5 mg
Drug: Progenta — 25 mg, administered as a once daily oral dose for 90 days.
  Other Names: CDB-4124; Telapristone acetate
  Arms: progenta 25 mg
Drug: Progenta — 50 mg, administered as a once daily oral dose for 90 days.
  Other Names: CDB-4124
  Arms: progenta 50 mg
Drug: Lucron Depot — 3.75 mg IM monthly
  Other Names: leuprolide acetate for depot suspension
  Arms: Lucron Depot
Drug: Placebo — Administered as a once daily oral dose for 90 days.
  Arms: placebo

SUMMARY:
A study of 3 doses of Progenta versus placebo versus Lucron Depot for treatment of leiomyomata.

DETAILED DESCRIPTION:
Three doses of Progenta (CDB4124 - 12.5, 25, 50 mg) versus placebo versus Lucron Depot (leuprolide acetate for depot suspension) was initiated in females with symptomatic leiomyomata. A single dose PK visit was conducted only for subjects randomized to the Progenta arm, between screening and visit 1. A second PK assessment was conducted at Visit 3 (one month on drug) to collect steady state data. Treatment period lasted for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Had at least one leiomyomata lesion that was identifiable and measurable by transvaginal ultrasound.
* Had a regular or steady menstrual cycle lasting from 24 to 36 days.

Exclusion Criteria:

* Post-menopausal
* Subject with documented endometriosis

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2004-07; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Assess the safety of Progenta when administered in pre-menopausal women with symptomatic leiomyomata. | 90 days

SECONDARY OUTCOMES:
Determine the tolerability of three doses of Progenta (12.5 mg, 25 mg, and 50 mg) as compared to placebo and Lucron Depot (leuprolide acetate for depot suspension) in pre-menopausal women with symptomatic leiomyomata. | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Wiehle, PhD, Study Director — Repros Therapeutics Inc.
Locations (1):
- Medical University /MTZ Clinical Research Sp.zo.o., Warsaw, Poland